CLINICAL TRIAL: NCT03629223
Title: Phase 1, Open-label, 3-Parts Study With Crossover Design in Each Part to Investigate the Bioequivalence of the Tablet Formulation of TF3 Compared to TF2 (Part A), and to Investigate the Influence of Food on the PK of Each TF2 (Part B) and TF3 (Part C) of Tepotinib in Healthy Subjects
Brief Title: Bioequivalence of TF3 and TF2 and Effect of Food on the PK of Tepotinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200095_0044; 2017-005056-29 (EudraCT Number)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: Tepotinib; Pharmacokinetics; Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A: First Tepotinib TF2 then TF3 (Experimental): Participants received a single oral dose of 500 milligrams (mg) Tepotinib tablet formulation 2 (TF2, reference treatment) on Day 1 of treatment period 1 followed by a single oral dose of 500 mg (2 x 250 mg) Tepotinib tablet formulation 3 (TF3, test treatment) on Day 1 of treatment period 2 under fasting conditions. The washout period was 21 days between Day 1 of each period.
  Interventions: Drug: Tepotinib TF2; Drug: Tepotinib TF3
- Part A: First Tepotinib TF3 then TF2 (Experimental): Participants received a single oral dose of 500 mg (2 x 250 mg) Tepotinib TF3 (test treatment) on Day 1 of treatment period 1 followed by a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of treatment period 2 under fasting conditions. The washout period was 21 days between Day 1 of each period.
  Interventions: Drug: Tepotinib TF2; Drug: Tepotinib TF3
- Part B: First Tepotinib TF2 Fasted then TF2 Fed (Experimental): Participants received a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of treatment period 1 under fasting conditions followed by a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of treatment period 2 under fed conditions. The washout period was 21 days between Day 1 of each period.
  Interventions: Drug: Tepotinib TF2
- Part B: First Tepotinib TF2 Fed then TF2 Fasted (Experimental): Participants received a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of treatment period 1 under fed conditions followed by a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of treatment period 2 under fasting conditions. The washout period was 21 days between Day 1 of each period.
  Interventions: Drug: Tepotinib TF2
- Part C: First Tepotinib TF3 Fasted then TF3 Fed (Experimental): Participants received a single oral dose of 500 mg (2 x 250 mg) Tepotinib TF3 (test treatment) on Day 1 of treatment period 1 under fasting conditions followed by a single oral dose of 500 mg (2 x 250 mg) Tepotinib TF3 (test treatment) on Day 1 of treatment period 2 under fed conditions. The washout period was 21 days between Day 1 of each period.
  Interventions: Drug: Tepotinib TF3
- Part C: First Tepotinib TF3 Fed then TF3 Fasted (Experimental): Participants received a single oral dose of 500 mg (2 x 250 mg) Tepotinib TF3 (test treatment) on Day 1 of treatment period 1 under fed conditions followed by a single oral dose of 500 mg (2 x 250 mg) Tepotinib TF3 (test treatment) on Day 1 of treatment period 2 under fasting conditions. The washout period was 21 days between Day 1 of each period.
  Interventions: Drug: Tepotinib TF3

INTERVENTIONS:
Drug: Tepotinib TF2 — Participants received a single oral dose of 500 mg Tepotinib TF2 under fasting or fed conditions in treatment period 1 or 2.
  Arms: Part A: First Tepotinib TF2 then TF3; Part A: First Tepotinib TF3 then TF2; Part B: First Tepotinib TF2 Fasted then TF2 Fed; Part B: First Tepotinib TF2 Fed then TF2 Fasted
Drug: Tepotinib TF3 — Participants received single oral dose of 500 mg (2 x 250 mg)Tepotinib TF3 under fasting or fed conditions in treatment period 1 or 2.
  Arms: Part A: First Tepotinib TF2 then TF3; Part A: First Tepotinib TF3 then TF2; Part C: First Tepotinib TF3 Fasted then TF3 Fed; Part C: First Tepotinib TF3 Fed then TF3 Fasted

SUMMARY:
The main purpose of the study was to demonstrate bioequivalence between the new tablet formulation (TF3, test treatment) and the tablet formulation used in clinical studies (TF2, reference treatment) and to investigate effect of food on pharmacokinetics (PK) of tepotinib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants of non-child bearing potential
* Body weight between 50 to 100 kilogram (kg)
* Body mass index (BMI) between 18.5 and 29.9 kilogram per meter square (kg/m^2)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participation in a clinical study within 60 days prior to first drug administration
* Whole blood donation or loss of greater than 450 milliliter (mL) within 60 days prior to first drug administration
* Any surgical or medical condition, or any other significant disease that could interfere with the study objectives, conduct, or evaluation
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0044
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 142 participants were screened in this study. Out of which 66 participants were randomized into the study.
Period: Treatment Period 1 (21 Days)
Arm/Group | Part A: First Tepotinib TF2 Then TF3 | Part A: First Tepotinib TF3 Then TF2 | Part B: First Tepotinib TF2 Fasted Then TF2 Fed | Part B: First Tepotinib TF2 Fed Then TF2 Fasted | Part C: First Tepotinib TF3 Fasted Then TF3 Fed | Part C: First Tepotinib TF3 Fed Then TF3 Fasted
Started | 20 | 20 | 6 | 8 | 6 | 6
Completed | 20 | 18 | 6 | 6 | 6 | 6
Not Completed | 0 | 2 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Benzodiazepines positive | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Toothache treatment | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (21 Days)
Arm/Group | Part A: First Tepotinib TF2 Then TF3 | Part A: First Tepotinib TF3 Then TF2 | Part B: First Tepotinib TF2 Fasted Then TF2 Fed | Part B: First Tepotinib TF2 Fed Then TF2 Fasted | Part C: First Tepotinib TF3 Fasted Then TF3 Fed | Part C: First Tepotinib TF3 Fed Then TF3 Fasted
Started | 20 | 18 | 6 | 6 | 6 | 6
Completed | 19 | 18 | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did not attend the ambulatory visits | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis set included all participants who had received at least 1 dose of planned study drug in the respective parts.
Groups:
- Part A: All Participants: All participants who received a single oral dose of 500 mg Tepotinib TF2 (reference treatment) (1*500 mg) or a single oral dose of Tepotinib TF3 (test treatment) (2*250 mg tablet) on Day 1 of either treatment period 1 or 2 under fasted conditions.
- Part B: All Participants: All participants who received a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of either treatment period 1 or 2 under fasted or fed conditions.
- Part C: All Participants: All participants who received a single oral dose of 500 mg (2 x 250 mg) Tepotinib TF3 (test treatment) on Day 1 of either treatment period 1 or 2 under fasted or fed conditions.
- Total: Total of all reporting groups
Arm/Group | Part A: All Participants | Part B: All Participants | Part C: All Participants | Total
Number analyzed (Participants) | 40 | 14 | 12 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 14 | 12 | 66
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 0 | 5
  Male | 36 | 13 | 12 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 39 | 14 | 12 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 38 | 14 | 12 | 64
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A, B and C: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable Concentration (AUC 0-t) of Tepotinib
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144 and 168 hours post-dose on Day 1 of each treatment period
Population: Pharmacokinetic.(PK) Analysis Set included participants without any relevant protocol deviations with respect to PK and absence of factors likely to affect comparability of PK results, with adequate trial medication compliance, who had valid primary endpoints for both treatments for Part A; and who had at least 3 post-dose concentration measurements for Part B; C.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Groups:
- Part A: TF2, Fasted: Participants received a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of either treatment period 1 or of treatment period 2 under fasting conditions.
- Part A: TF3, Fasted; Part C: TF3, Fasted: Participants received a single oral dose of 500 mg (2 x 250 mg) Tepotinib TF3 (test treatment) on Day 1 of either treatment period 1 or treatment period 2 under fasting conditions.
- Part B: TF2, Fasted: Participants received a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of either treatment period 1 or treatment period 2 under fasting conditions.
- Part B: TF2, Fed: Participants received a single oral dose of 500 mg Tepotinib TF2 (reference treatment) on Day 1 of either treatment period 1 or treatment period 2 under fed conditions.
- Part C: TF3, Fed: Participants received a single oral dose of 500 mg (2 x 250 mg) Tepotinib TF3 (test treatment) on Day 1 of either treatment period 1 or treatment period 2 under fed conditions.
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 38 | 12 | 14 | 12 | 12
nanograms*hour per milliliter (ng*h/mL) | 16146 (23.4) | 18645 (21.0) | 12609 (38.1) | 23457 (25.1) | 17964 (19.8) | 29307 (25.0)
Statistical Analysis 1: Comparison: Part A: TF2, Fasted vs Part A: TF3, Fasted; Test type: Equivalence — Analysis was performed with Equivalence acceptance range for 90% confidence interval (CI) as 80.00% - 125.00%. In the below, LS-means = least squares mean; Percentage of Ratio of Geometric LS-Mean = 115.35, 90% CI 2-sided [108.55 to 122.58]
Statistical Analysis 2: Comparison: Part B: TF2, Fasted vs Part B: TF2, Fed; Test type: Other; Percentage of ratio of Geometric LS-Mean = 186.37, 90% CI 2-sided [163.61 to 212.28]
Statistical Analysis 3: Comparison: Part C: TF3, Fasted vs Part C: TF3, Fed; Test type: Other; Percentage of ratio of Geometric LS-Mean = 163.15, 90% CI 2-sided [146.17 to 182.10]

2. Primary Outcome: Part A, B and C: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC 0-inf) of Tepotinib
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/ lambda z, where Clast is the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and lambda z is the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: as for outcome 1
Population: PK Analysis Set included participants without any relevant protocol deviations with respect to PK and absence of factors likely to affect comparability of PK results, with adequate trial medication compliance, who had valid primary endpoints for both treatments for Part A; and who had at least 3 post-dose concentration measurements for Part B; C.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 38 | 12 | 14 | 12 | 12
ng*h/mL | 16728 (23.9) | 19316 (21.3) | 13037 (38.2) | 24443 (25.9) | 18447 (20.0) | 30118 (25.5)
Statistical Analysis 1: Comparison: Part A: TF2, Fasted vs Part A: TF3, Fasted; Test type: Equivalence — Analysis was performed with Equivalence acceptance range for 90% confidence interval (CI) as 80.00% - 125.00%; Percentage of ratio of Geometric LS-Mean = 115.34, 90% CI 2-sided [108.51 to 122.60]
Statistical Analysis 2: Comparison: Part B: TF2, Fasted vs Part B: TF2, Fed; Test type: Other; Percentage of ratio of Geometric LS-Mean = 186.67, 90% CI 2-sided [163.78 to 212.77]
Statistical Analysis 3: Comparison: Part C: TF3, Fasted vs Part C: TF3, Fed; Test type: Other; Percentage of ratio of Geometric LS-Mean = 163.26, 90% CI 2-sided [146.09 to 182.46]

3. Primary Outcome: Part A, B and C: Maximum Observed Plasma Concentration (Cmax) of Tepotinib
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 38 | 12 | 14 | 12 | 12
ng/mL | 253 (20.6) | 288 (22.5) | 199 (29.5) | 476 (19.6) | 280 (15.3) | 559 (17.0)
Statistical Analysis 1: Comparison: Part A: TF2, Fasted vs Part A: TF3, Fasted; Test type: Equivalence — Analysis was performed with equivalence acceptance range for 90% confidence interval (CI) as 80.00% - 125.00%; Percentage of ratio of Geometric LS-Mean = 113.57, 90% CI 2-sided [107.62 to 119.85]
Statistical Analysis 2: Comparison: Part B: TF2, Fasted vs Part B: TF2, Fed; Test type: Other; Percentage of ratio of Geometric LS-Mean = 236.51, 90% CI 2-sided [215.69 to 259.34]
Statistical Analysis 3: Comparison: Part C: TF3, Fasted vs Part C: TF3, Fed; Test type: Other; Percentage of ratio of Geometric LS-Mean = 199.61, 90% CI 2-sided [176.44 to 225.82]

4. Secondary Outcome: Part A, B and C: Time to Reach the Maximum Plasma Concentration (Tmax) of Tepotinib
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 38 | 12 | 14 | 12 | 12
hours | 14.1 [6.00 to 48.0] | 12.0 [8.00 to 36.0] | 24.0 [6.00 to 48.0] | 12.0 [4.00 to 12.0] | 12.0 [3.00 to 36.0] | 8.0 [6.00 to 12.0]

5. Secondary Outcome: Part A, B and C: Terminal Half-Life (t1/2) of Tepotinib
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z. Lambda z is the terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 38 | 12 | 14 | 12 | 12
hours | 31.8 (17.8) | 30.9 (15.3) | 30.8 (11.6) | 30.0 (12.9) | 29.2 (14.7) | 29.9 (14.5)

6. Secondary Outcome: Part A, B and C: Apparent Total Body Clearance of Tepotinib From Plasma Following Oral Administration (CL/f)
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 38 | 12 | 14 | 12 | 12
liter per hour | 26.9 (23.9) | 23.3 (21.3) | 34.5 (38.2) | 18.4 (25.9) | 24.4 (20.0) | 14.9 (25.5)

7. Secondary Outcome: Part A, B and C: Apparent Volume of Distribution of Tepotinib During the Terminal Phase Following Extravascular Administration (Vz/f)
Description: Vz/f was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) is influenced by the fraction absorbed and was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/f after oral dose is influenced by the fraction absorbed.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 38 | 12 | 14 | 12 | 12
liter | 1232 (28.5) | 1038 (24.3) | 1531 (40.8) | 797 (27.0) | 1027 (24.9) | 644 (26.3)

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: Time from date of informed consent signature up to end of study (assessed up to 7 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 40 | 12 | 14 | 12 | 12
Participants
  Participants with TEAEs | 18 | 14 | 5 | 9 | 6 | 6
  Participants with Serious TEAEs | 0 | 0 | 0 | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Values
Description: The laboratory measurements included hematology, blood chemistry and urinalysis. Number of participants with clinically significant abnormalities in laboratory values were reported. Clinically Significance was decided by investigator.
Time Frame: Time from date of informed consent signature up to end of study (assessed up to 7 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 40 | 12 | 14 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG) Findings
Description: The 12-lead ECG recordings were obtained after 5 minutes of rest in a semi-supine position. ECG recordings included rhythm, ventricular rate, PR interval, QRS duration, QT and QTc intervals. Number of participants with clinically significant abnormalities in 12-lead ECG findings were reported. Clinically significance was decided by investigator.
Time Frame: Time from date of informed consent signature up to end of study (assessed up to 7 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 40 | 12 | 14 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital sign assessment included blood pressure, pulse rate and body temperature. Number of participants with clinically significant abnormalities in vital signs were reported. Clinically significance was decided by investigator.
Time Frame: Time from date of informed consent signature up to end of study (assessed up to 7 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
Number analyzed (Participants) | 38 | 40 | 12 | 14 | 12 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Time from date of informed consent signature up to end of study (assessed up to 7 weeks)
Description: The Safety analysis set included all participants who had received at least 1 dose of planned study drug in the respective parts.
Arm/Group | Part A: TF2, Fasted | Part A: TF3, Fasted | Part B: TF2, Fasted | Part B: TF2, Fed | Part C: TF3, Fasted | Part C: TF3, Fed
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40 | 0/12 | 0/14 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40 | 0/12 | 1/14 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 18/38 | 14/40 | 5/12 | 9/14 | 6/12 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: TF2, Fasted (N=38) | Part A: TF3, Fasted (N=40) | Part B: TF2, Fasted (N=12) | Part B: TF2, Fed (N=14) | Part C: TF3, Fasted (N=12) | Part C: TF3, Fed (N=12)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: TF2, Fasted (N=38) | Part A: TF3, Fasted (N=40) | Part B: TF2, Fasted (N=12) | Part B: TF2, Fed (N=14) | Part C: TF3, Fasted (N=12) | Part C: TF3, Fed (N=12)
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0 | 2 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 | 5 | 1 | 3 | 5 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 2
Radisectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT03629223/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT03629223/SAP_001.pdf